CLINICAL TRIAL: NCT03105661
Title: Use of Impedance Cardiography to Decrease the Risk of Preeclampsia in Obese Patients
Brief Title: Use of Impedance Cardiography to Decrease the Risk of Pre-eclampsia in Obese Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Mary Ellen McNeal, Research Coordinator, University of Tennessee Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4226
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Obesity, Morbid; Preeclampsia
MeSH Terms: conditions — Obesity, Morbid; Pre-Eclampsia | interventions — Labetalol; Nifedipine; Atenolol

STUDY DESIGN:
Intervention Model Description: Randomization to treatment or non treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm (Active Comparator): Patients will be randomized to treatment with antihypertensive medications used with pregnancy for thirty years.
  Labetalol Hydrochloride 200 mg orally every 12 hours Nifedipine 60 mg orally daily Atenolol 25 mg daily
  Interventions: Drug: Labetalol Hydrochloride 200 mg; Drug: NIFEdipine 60 mg; Drug: Atenolol 25 mg
- Non-treatment Arm (No Intervention): Patients who are randomized to the non-treatment arm will not receive antihypertensive medications.

INTERVENTIONS:
Drug: Labetalol Hydrochloride 200 mg — Anti-hypertensive prescribed for increased cardiac output as determined by Impedance Cardiography
  Other Names: Trandate
  Arms: Treatment Arm
Drug: NIFEdipine 60 mg — Anti-hypertensive medication prescribed for increased systemic vascular resistance as determined by Impedance Cardiography
  Other Names: Procardia
  Arms: Treatment Arm
Drug: Atenolol 25 mg — Anti-hypertensive prescribed for increased cardiac output with tachycardia or maternal pulse rate 110 or greater
  Other Names: Tenormin
  Arms: Treatment Arm

SUMMARY:
To determine if the use of impedance cardiography can identify appropriate medications for use in treating morbidly obese patients to decrease the risk of preeclampsia.

DETAILED DESCRIPTION:
Research Protocol

Use of Impedance Cardiography to decrease the risk of preeclampsia in obese patients

Background: Obesity is epidemic in the United States and this is leading to an increase in the number of pregnant patients with obesity. Obesity, especially morbid obesity (BMI >/= 40), increases the risk of developing preeclampsia when compared to the non-obese population. Impedance Cardiography has never been used to evaluate this patient population to see if they have abnormal cardiac output and/or abnormal peripheral resistance. If identified, low dose medical treatment can be done to normalize these patterns early on to see if this treatment modality decreases the development of preeclampsia and other pregnancy complications.

Specific Aims: The primary aim of this study is to determine if the use of Impedance Cardiography can help identify the appropriate medicine for use in treating morbidly obese patients that have abnormal testing results, to see if by normalizing impedance cardiography testing parameters results in a decrease in the incidence of preeclampsia in general and other pregnancy complications.

Enrollment: All pregnant patients, 18-51 years old, less than 20 weeks pregnant, with a BMI >/= 40 will undergo impedance cardiography and if the results are abnormal, will be provided informed consent to participate. If consent is given, and blood pressure is < 140/90,they will be eligible for enrollment.

Randomization: All patients who meet criteria will undergo impedance cardiography. Those with abnormal results will be randomized as the whether they will be treated or not. Randomization will require they blindly pull a paper labelled "yes" or "no" from a container. Those who select "yes" will be randomized to the treatment arm and will be prescribed antihypertensive medications commonly used in obstetrics for hypertension (labetalol, nifedipine, atenolol) Those who select "no" will not receive medication.

Study Procedure: All pregnant patients that meet study criteria and have abnormal Impedance Cardiography testing will be asked to participate, consented and randomized to the treatment or non treatment arm. The treatment group will receive antihypertensive medications as listed above and undergo monthly cardiography testing after beginning treatment with medication adjustments until normal test results are obtained. The non treatment group will undergo repeat cardiography testing 8 weeks after the first test to compare results. All enrolled patients will be followed with regular prenatal care for their prospective conditions and followed closely for the development of high or low blood pressure and preeclampsia.

Adverse events: Adverse events related to this study are minimal because the test is non invasive and complications for Impedance Cardiology are non existent. In addition, the drugs used to treat hypertension have been used in obstetrics for over 30 years with good results and minimal problems.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients 18-51 years old,
* Less than 20 weeks gestation with Morbid Obesity (BMI >/= 40)
* Not on antihypertensive medications

Exclusion Criteria:

* Patients with an allergy to antihypertensive medication or contraindication for their usage such as certain cardiac or neurologic disorder during pregnancy
* Patients who have a blood pressure 140/90 or greater

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-04 (Estimated)

PRIMARY OUTCOMES:
Rates of preeclampsia in morbidly obese pregnant women | 2 years
  Rates of preeclampsia in morbidly obese pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Craig V. Towers, MD, Principal Investigator — University of Tennessee Graduate School of Medicine
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No